CLINICAL TRIAL: NCT03357536
Title: Genetic Susceptibility to Listeriosis - Listeria-GEN
Brief Title: Genetic Susceptibility to Listeriosis
Acronym: Listeria-GEN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2014-31; ID-RCB number : 2015-A01386-43 (Other: French national registration number of the study)
Record Dates: First submitted 2017-11-24; First posted 2017-11-30 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Listeriosis
MeSH Terms: conditions — Listeriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with Listeriosis (Experimental): Patients with Listeriosis.
  Human biological samples :
  * Blood sample
  * Skin biopsy
  * Saliva
  Interventions: Procedure: Human biological samples
- Volunteers related with patients with Listeriosis (Experimental): Volunteers related with patients with Listeriosis.
  Human biological samples :
  * Blood sample
  * Skin biopsy
  * Saliva
  Interventions: Procedure: Human biological samples

INTERVENTIONS:
Procedure: Human biological samples — * Blood sample
  * Skin biopsy
  * Saliva

SUMMARY:
Listeriosis is a rare, severe foodborne infection, responsible for severe invasive infections. It occurs in the great majority of cases in elderly patients and / or patients with comorbidities, with a deficit of innate or cellular immunity. Pregnancy is also a risk factor.

The Multicentric Observational NAtional Analysis of Listeriosis and Listeria (MONALISA) is an ongoing national case-control prospective study on listeriosis implemented since 2009 to study risk and prognosis factors for listeriosis. In this cohort, which enrolled 902 patients on 1 August 2014, 7% of patients with neurolisteriosis are under 40 years of age and have no identified risk factor. Genetic susceptibility is suspected in these patients. Genetic susceptibility could also explain the inconstant development of a neurolisteriosis or fetal infection, as well as the particular severity of some infections (death, foetal loss, neurological sequelae).

The aim of the study is to identify genetic susceptibility to Listeriosis.

DETAILED DESCRIPTION:
Listeriosis is a rare, severe foodborne infection caused by the bacterium Listeria monocytogenes (Lm), responsible for severe invasive infections. It occurs in the great majority of cases in elderly patients and / or patients with comorbidities, with a deficit of innate or cellular immunity. Pregnancy is also a risk factor.

The Multicentric Observational NAtional Analysis of Listeriosis and Listeria (MONALISA) is an ongoing national case-control prospective study on listeriosis implemented since 2009 to study risk and prognosis factors for listeriosis. In this cohort, which enrolled 902 patients on 1 August 2014, 7% of patients with neurolisteriosis are under 40 years of age and have no identified risk factor. Genetic susceptibility is suspected in these patients. Genetic susceptibility could also explain the inconstant development of a neurolisteriosis or fetal infection, as well as the particular severity of some infections (death, foetal loss, neurological sequelae).

The analysis of the genetically transmitted vulnerability of Lm has not yet been studied, because of the lack of accessibility to prospective cohorts (and their DNA) for this rare and severe infection.

The aim of the study is to identify genetic susceptibility to Listeriosis that will optimize the patient care in terms of treatment and prevention.

ELIGIBILITY:
Inclusion Criteria for patients with Listeriosis :

* Microbiologically documented Listeriosis (either a severe form of listeriosis, or an atypical form of listeriosis, or less than 40 years old and without any co-morbidity identified)
* Affiliated or beneficiary of a social security system
* Informed and written consent

Inclusion Criteria for volunteers related to patients with Listeriosis (after identifying a genetic susceptibility in the patient with Listeriosis) :

* defined as father, mother, brother (s), sister (s), child (ren), grandparent (s), uncle (s), aunt (s), cousin (s), nephew (s), niece (s).
* Affiliated or beneficiary of a social security system
* Informed and written consent

Exclusion Criteria for volunteers related to patients with Listeriosis:

* Inability to consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-11-28 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Identification of a susceptibility factor associated with Listeriosis infection | 10 years
  In patients with Listeriosis, the hypothesis that the identified genetic variation is the mutation responsible for the infection will be verified :
  * by verifying that it is not a listed polymorphism by sequencing genomic DNA controls
  * by verifiyng that family genetic segregation is compatible with clinical segregation
  * by verifying the function of the mutated protein in the patient's cell lines and / or fresh cells
  * by performing complementation experiments by transfecting the wild-type allele into the patient's cells

SECONDARY OUTCOMES:
Identification of a susceptibility factor associated with the most severe or atypical forms | 10 years
  In patients with Listeriosis, the susceptibility factor associated with the most severe or atypical forms will be characterized :
  * By testing the response and production of cytokines involved in infection control.
  * By identifying chromosomal regions associated with the disease by a homozygosity mapping genetic study on multiplex and / or inbred families.
  * By sequencing the identified candidate genes.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Lecuit, Study Director — Institut Pasteur
Locations (1):
- Centre Médical de l'Institut Pasteur, Paris, France

IPD SHARING:
Plan to Share IPD: No